CLINICAL TRIAL: NCT00657514
Title: Evaluation of Ranolazine on Skeletal Muscle Endpoints During Exercise In Subjects With Chronic Angina and Peripheral Arterial Disease
Brief Title: Ranolazine Versus Placebo Effects on Exercise Tolerance in Patients With Heart Disease and Peripheral Arterial Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Colorado Prevention Center (Other)
Responsible Party: Principal Investigator, Mark Nehler, MD, Chief, Section of Vascular Surgery and EndoVascular Therapy and Podiatry, Colorado Prevention Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-PAD-01
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Peripheral Arterial Disease; Angina
Keywords: hemoglobin desaturation kinetics; peripheral arterial disease; chronic angina; exercise tolerance
MeSH Terms: conditions — Peripheral Arterial Disease; Angina Pectoris | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Drug arm - 500mg tablet po bid up to 1000mg (2 500mg tablets) po bid
  Interventions: Drug: Ranolazine
- P (Placebo Comparator): Placebo arm - 1 tablet po bid up to 2 tablets po bid if tolerated
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 500mg tablet po bid up to 1000mg (2 500mg tablets) po bid
  Other Names: Ranexa, extended-release tablets; CVT500; light orange; NDC Code: 67159-112-04
  Arms: A
Drug: Placebo — 1 tablet po bid up to 2 tablets po bid if tolerated
  Arms: P

SUMMARY:
After 6 weeks of maximal Ranolazine therapy, tissue hemoglobin desaturation kinetics will change compared to placebo in patients with chronic angina and peripheral arterial disease.

DETAILED DESCRIPTION:
Study Endpoints:

Primary Endpoint:

• The primary endpoint of this study is the change in the kinetics of tissue hemoglobin oxygen desaturation (expressed as time constants) following the onset of exercise.

Secondary endpoints of this study include percent and absolute change in:

* Peak oxygen consumption
* Pulmonary oxygen uptake on-kinetics
* Steady state level of tissue hemoglobin desaturation during exercise
* Recovery kinetics of tissue oxygen saturation following exercise

Adverse events will be collected.

Exploratory Endpoints

* Peak Walking Time (PWT)
* Claudication Onset Time (COT)
* Time to Onset of Angina (TOA)

Study Design:

Investigator-initiated, prospective, randomized, double-blind, placebo-controlled study.

Inclusion Criteria:

1. Males age > 40 years.
2. Subjects must have chronic stable angina, meeting the labeled indications for ranolazine:

   • Ranolazine is indicated for the treatment of chronic angina. Ranolazine should be reserved for subjects who have not achieved an adequate response with other anti-anginal drugs.
3. Subjects must have a resting ankle brachial index (ABI) of < 0.90 with a post-exercise decrement of ≥ 10% in at least one leg, OR a resting ABI of ≥0.90 to ≤ 1.00 with a post-exercise decrement of ≥ 20% in at least one leg
4. The subject has provided written informed consent to participate, understands the requirements of the study, and agrees to return for the required assessments

Exclusion Criteria:

1. Non-atherosclerotic diseases of the peripheral circulation by clinical history
2. Unable to complete the first stage of the modified, extended Astrand treadmill protocol
3. Clinically significant ECG abnormalities or changes with exercise on the screening ECG
4. Evidence of critical limb ischemia (CLI)
5. Hepatic impairment (Child-Pugh Classes A [mild], B [moderate], or C [severe])
6. End stage renal disease requiring dialysis
7. Hemoglobin < 12 mg/dL.
8. Platelet count < 90,000/mL.
9. Planned surgical/endovascular intervention for coronary artery disease (CAD) or peripheral arterial disease (PAD) in the next 3 months
10. Maximal exercise is limited by symptoms other than claudication or angina
11. Significant mental illness or drug abuse within 30 days of enrollment that in the opinion of the Investigator could impact the subject's ability to successfully complete the trial
12. Known allergy to ranolazine
13. Pre-existing QTc prolongation on a resting electrocardiogram (ECG) at Screening due to the risk of worsening of this condition with the use of ranolazine
14. Treatment with QT prolonging drugs such as Class IA (e.g. quinidine) and Class III (e.g. sotalol, dofetilide), antiarrhythmics, amiodarone, and antipsychotics (e.g. thioridazine, ziprasidone)
15. Treatment with potent or moderately potent CYP3A inhibitors including ketoconazole and other azole antifungals, diltiazem, verapamil, macrolide antibiotics, cyclosporine, rifampin or structurally related rifabutin and rifapentin, phenobarbital, phenytoin, carbamazepine, St. John's Wort, or human immunodeficiency virus (HIV) protease inhibitors
16. The subject has previously received ranolazine within the 6-months prior to enrollment
17. The subject has received an investigational drug within 90 days prior to enrollment
18. Type 1 or type 2 diabetes mellitus
19. Congestive Heart Failure, ≥ New York Heart Association (NYHA) Class III
20. History of oxygen dependent Chronic Obstructive Pulmonary Disease (COPD)
21. Body Mass Index (BMI) >35

ELIGIBILITY:
Inclusion Criteria:

* Males age > 40 years.
* Subjects must have chronic stable angina, meeting the labeled indications for ranolazine:

Ranolazine is indicated for the treatment of chronic angina. Ranolazine should be reserved for subjects who have not achieved an adequate response with other anti-anginal drugs.

* Subjects must have a resting ankle brachial index (ABI) of < 0.90 with a post-exercise decrement of ≥ 10% in at least one leg, OR a resting ABI of ≥0.90 to ≤ 1.00 with a post-exercise decrement of ≥ 20% in at least one leg
* The subject has provided written informed consent to participate, understands the requirements of the study, and agrees to return for the required assessments

Exclusion Criteria:

* Non-atherosclerotic diseases of the peripheral circulation by clinical history
* Unable to complete the first stage of the modified, extended Astrand treadmill protocol
* Clinically significant ECG abnormalities or changes with exercise on the screening ECG
* Evidence of critical limb ischemia (CLI)
* Hepatic impairment (Child-Pugh Classes A [mild], B [moderate], or C [severe])
* End stage renal disease requiring dialysis
* Hemoglobin < 12 mg/dL.
* Platelet count < 90,000/mL.
* Planned surgical/endovascular intervention for coronary artery disease (CAD) or peripheral arterial disease (PAD) in the next 3 months
* Maximal exercise is limited by symptoms other than claudication or angina
* Significant mental illness or drug abuse within 30 days of enrollment that in the opinion of the Investigator could impact the subject's ability to successfully complete the trial
* Known allergy to ranolazine
* Pre-existing QTc prolongation on a resting electrocardiogram (ECG) at Screening due to the risk of worsening of this condition with the use of ranolazine
* Treatment with QT prolonging drugs such as Class IA (e.g. quinidine) and Class III (e.g. sotalol, dofetilide), antiarrhythmics, amiodarone, and antipsychotics (e.g. thioridazine, ziprasidone)
* Treatment with potent or moderately potent CYP3A inhibitors including ketoconazole and other azole antifungals, diltiazem, verapamil, macrolide antibiotics, cyclosporine, or human immunodeficiency virus (HIV) protease inhibitors
* The subject has previously received ranolazine within the 6-months prior to enrollment
* The subject has received an investigational drug within 90 days prior to enrollment
* Type 1 or type 2 diabetes mellitus
* Congestive Heart Failure, ≥ New York Heart Association (NYHA) Class III
* History of oxygen dependent Chronic Obstructive Pulmonary Disease (COPD)
* Body Mass Index (BMI) >35

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
skeletal muscle hemoglobin desaturation kinetics | 6 weeks

SECONDARY OUTCOMES:
peak exercise oxygen consumption | 6 weeks
Pulmonary oxygen uptake on-kinetics | 6 weeks
Steady state level of tissue hemoglobin desaturation during exercise | 6 weeks
Recovery kinetics of tissue oxygen saturation following exercise | 6 weeks
adverse events | 6 weeks
Peak Walking Time (PWT) | 6 weeks
Claudication Onset Time (COT) | 6 weeks
Time to Onset of Angina (TOA) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Nehler, MD, Principal Investigator — The Univesity of Colorado at Denver; William R Hiatt, MD, Study Chair — Colorado Prevention Center
Locations (3):
- United States (3):
  - University of Colorado at Denver, Aurora, Colorado
  - Denver Health and Hospital Authority (DHHA), Denver, Colorado
  - Department of Veteran Affairs Medical Center, Denver, Colorado

REFERENCES:
- [Background] Bauer TA, Regensteiner JG, Brass EP, Hiatt WR. Oxygen uptake kinetics during exercise are slowed in patients with peripheral arterial disease. J Appl Physiol (1985). 1999 Aug;87(2):809-16. doi: 10.1152/jappl.1999.87.2.809. PMID 10444643
- [Background] Barstow TJ, Lamarra N, Whipp BJ. Modulation of muscle and pulmonary O2 uptakes by circulatory dynamics during exercise. J Appl Physiol (1985). 1990 Mar;68(3):979-89. doi: 10.1152/jappl.1990.68.3.979. PMID 2341363
- [Background] Bauer TA, Brass EP, Hiatt WR. Impaired muscle oxygen use at onset of exercise in peripheral arterial disease. J Vasc Surg. 2004 Sep;40(3):488-93. doi: 10.1016/j.jvs.2004.06.025. PMID 15337878